CLINICAL TRIAL: NCT02877381
Title: Tranexamic Acid in Revision Total Joint Arthroplasty: A Prospective Randomized Controlled Trial
Brief Title: Tranexamic Acid in Revision Total Joint Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Chief of Adult Reconstruction, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15063007
Record Dates: First submitted 2016-04-14; First posted 2016-08-24 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Revision Total Knee Arthroplasty; Revision Total Hip Arthroplasty; Acute Blood Loss Anemia
Keywords: Tranexamic Acid; Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single IV Dose (Active Comparator): • 1 gram IV TXA administered at time of prepping and draping
  Interventions: Procedure: Revision Total Knee Arthroplasty (TKA); Procedure: Revision Total Hip Arthroplasty (THA)
- Double Dose IV (Active Comparator): * 1 gram IV TXA administered at time of prepping and draping
  * 1 gram IV TXA administered prior to tourniquet deflation
  Interventions: Procedure: Revision Total Knee Arthroplasty (TKA); Procedure: Revision Total Hip Arthroplasty (THA)
- IV + Topical (Active Comparator): * 1 gram IV TXA administered at time of prepping and draping
  * 1 gram topical TXA injected intra-articular following closure of the arthrotomy
  Interventions: Procedure: Revision Total Knee Arthroplasty (TKA); Procedure: Revision Total Hip Arthroplasty (THA)
- Repeated Oral Dose (Active Comparator): • Three 650 mg tablets of TXA administered two hours prior surgery with a second dose given 6 hours postoperatively and a final dose given the morning of postoperative day 1
  Interventions: Procedure: Revision Total Knee Arthroplasty (TKA); Procedure: Revision Total Hip Arthroplasty (THA)

INTERVENTIONS:
Procedure: Revision Total Knee Arthroplasty (TKA) — Femoral component exchange, tibial component exchange, both component exchange, explant of both components and placement of antibiotic cement spacer, or a second stage re-implantation procedure. Given the variability in blood loss between types of revision TKA, randomization will be done to ensure equivalent numbers of each type of revision TKA between the treatment groups.
Procedure: Revision Total Hip Arthroplasty (THA) — Femoral component exchange, acetabulum component exchange, both component exchange, explant of both components and placement of antibiotic cement spacer, or a second stage re-implantation procedure. Given the variability in blood loss between types of revision THA, randomization will be done to ensure equivalent numbers of each type of revision THA between the treatment groups.

SUMMARY:
To determine the optimal dosing regimen and route of administration of tranexamic acid (TXA) [single dose intravenous (IV), double dose intravenous, intravenous + topical, and oral repeated dosing] to minimize post-operative blood loss and transfusion requirements following revision total knee arthroplasty (RTKA).

DETAILED DESCRIPTION:
Study Design: Prospective randomized control study

Scientific Background/Intro: Total hip or knee arthroplasty is associated with the risk of moderate to significant blood loss. Approximately one-third of patients undergoing total joint replacement surgery require one to three units of blood postoperatively. Tranexamic acid is a synthetic antifibrinolytic agent that has been successfully used orally, intravenously, and topically to control bleeding after total joint replacement. The use of TXA has been shown to significantly reduce the need for blood products during total joint replacement.1-3

Many studies have explored the use of various TXA regimens following primary TKA. Tanaka et al. demonstrated both that pre-operative administration of TXA was superior to intra-operative administration and that a double dose regimen is superior to a single dose regimen.4 Maniar et al. further supported the idea that pre-operative TXA administration is superior, and the addition of higher doses of TXA improved efficacy without an increase in thromboembolic complications.5 More recently, Lin et al. demonstrated that combining a pre-operative IV dose of TXA with an intra-articular dose after arthrotomy closure was superior to an intra-articular dose alone.6 Also, in an unpublished randomized control trial that we recently completed, we found oral TXA to provide equivalent blood control at a lower cost than IV TXA.

It is well known that revision joint arthroplasty cases are more complex than primary joint replacements. Revision total knee arthroplasty is associated with a greater risk of blood loss and increased transfusion rates compared to primary TKA.7 Despite the vast body of literature investigating TXA following primary TKA, only three retrospective studies have been published on the use of TXA after revision TKA.8-10 All three studies have shown that IV TXA decreased both the rate of transfusions and the amount of blood transfused when compared to controls.8-10

Although the TXA formulations used in primary TKA have been shown to be effective in the retrospective studies, the amount of blood loss and risk of transfusion still remains significantly higher than during primary TKA. By performing the first randomized control trial on the use of TXA following revision TKA, we believe it will help change practice patterns by providing evidence that the same TXA formulations used in primary TKA are inadequate for revision TKA. Additionally, we will be exploring new combinations of TXA administration to answer some questions brought up by previous studies in regards to the optimal TXA regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for revision THA or TKA defined as femoral component exchange, acetabulum/tibial component exchange, both component exchange, explant of both components and placement of antibiotic cement spacer, or a second stage re-implantation procedure.

Exclusion Criteria:

* Patients scheduled for a head and liner/poly exchange, known allergy to TXA, acquired disturbances of color vision, refusal of blood products, pre-operative use of anticoagulant therapy within five days before surgery, a history of arterial or venous thrombotic disease (including a history of Deep Vein Thrombosis (DVT), Pulmonary Embolism (PE), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA)), pregnancy, breastfeeding, or major co-morbidities (myocardial infarction or stent placement within one year, severe pulmonary disease, renal impairment, or hepatic failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-04; Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Post-operative reduction in Hemoglobin | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Pre-operative hemoglobin minus the lowest post-operative hemoglobin prior to any transfusion
Post-operative reduction in Hematocrit | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Pre-operative hematocrit minus the lowest post-operative hematocrit prior to any transfusion
Calculated blood loss | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Based on predicted blood volume and hemoglobin balance
Number of units transfused | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  per patient
Number of Patients Transfused | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery

SECONDARY OUTCOMES:
Cost-comparison | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Cost differences resulted from differences in the blood transfusion rate, length of hospital stay, and management of complications as well as from the cost of the TXA itself
Deep Vein Thrombosis, Pulmonary Embolus, Cerebrovascular accident or Transient ischemic attack | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
Return to the OR within 30 days; Re-admission within 30 days; Periprosthetic fracture within 30 days | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
Superficial infection or Deep infection, defined as Synovial White Blood Cell (WBC) count > 4200 WBC/ml or Synovial WBC > 3000 WBC/ml & C-Reactive Protein (CRP) > 10 mg/dl & Erythrocyte Sedimentation Rate (ESR) > 30 mm/hr ; | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - New York University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided